CLINICAL TRIAL: NCT03246945
Title: Assessing Parental Photographs of Skin Disease and the Concordance of a Virtual Diagnosis: Can 3 Simple Instructions Improve Photograph Quality?
Brief Title: Photograph Quality Rating Scale Study ("PQRS Study")
Acronym: PQRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 15-012463
Record Dates: First submitted 2017-07-25; First posted 2017-08-11 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Dermatology/Skin - Other

STUDY DESIGN:
Intervention Model Description: Patient/parent dyads visiting a pediatric dermatology clinic were invited to participate. After consent, patient/parent dyads were randomly assigned to photography instruction versus no instruction. In both arms, parents photographed their child's skin condition (via smart phone) and provided medical history. Images were uploaded securely to the child's electronic health record for independent diagnosis by a dermatologist not involved in the patient's care.
Who Masked: Care Provider, Investigator
Masking Description: Dermatologist providing remote diagnosis was blinded to whether parents were provided instructions, which phone they took and the diagnosis provided by the in-person dermatologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): Patient-Parent Dyad receiving photography instructions prior to taking photographs of skin conditions
  Interventions: Behavioral: Instructions on taking photographs provided, see methods
- Control Arm (No Intervention): Patient-Parent Dyad not receiving photography instructions prior to taking photographs of skin conditions

INTERVENTIONS:
Behavioral: Instructions on taking photographs provided, see methods — Parent-patient dyads were provided with written 3-step instructions on how best to take a photograph of skin conditions using a smart phone
  Arms: Study Arm

SUMMARY:
Advances in smart phone-based photography (both quality and image transmission) offer the potential to greatly improve access to pediatric dermatologists. However, the accuracy of diagnoses reliant on parent-provided photographs has been neither measured nor compared to diagnoses based on in-person examinations. Therefore, the primary objective of this study was to assess the concordance between diagnoses based on photographs taken by parents (or legal guardians) and those based on in-person examinations. A secondary aim was to assess the effect of photography instructions on improving this concordance.

DETAILED DESCRIPTION:
Each patient/parent dyad will be randomized into one of two approximately equally sized groups; half of the subjects will be provided with an instruction sheet on how best to take photographs of skin conditions with their mobile devices (study group) and half will not be provided this instruction sheet (control group). Photographs will be evaluated for image quality and to provide a diagnosis (See attached forms including Photograph Quality Rating Scale).

ELIGIBILITY:
Inclusion Criteria:

1. Must be a new patient/parent dyad arrived at the main pediatric dermatology clinic
2. Patient must be under the age of 18.
3. Consenting parent or guardian must be present and able to speak English to participate.
4. Patients are either already enrolled in MyCHOP (MyChart) or are willing to enroll during the encounter.
5. Parent or legal guardian has a mobile phone with the capability to download the free MyChart app.
6. Parents have a data plan that allows them to download the MyChart app (if not already downloaded) and upload pictures, and are willing to accept any potential data charges incurred with these activities.
7. Patient has active skin lesion or rash that can be photographed during the clinic visit.

Exclusion Criteria:

1. Patient is over the age of 18.
2. Parent or guardian is not present or not able to speak English.
3. Parent or guardian is not able to enroll in MyCHOP (MyChart).
4. Parent or guardian does not have a mobile phone capable of downloading the MyChart app.
5. Photographs are not able to be taken (phone battery dies, phone/app does not work, patient is not cooperative, participant does not have time).
6. If there are no active skin lesions to photograph the patient/parent will not be enrolled (e.g. hives that are inactive, hyperhidrosis [excessive sweating], itching without a rash, resolved skin lesions [e.g. warts, molluscum]).
7. Patients presenting for a general full body skin exam will be excluded, as this would require full body photography, which is too time consuming. (Note: this does not include evaluation of one individual mole [nevus], which can be included in the study).

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The effect of photography instructions on average image quality, as evaluated using a photograph quality rating scale (PQRS) | 1 hour
  The PQRS quantifies photograph quality based on five criteria: clarity, perspective, darkness, brightness, and color. Each criterion is rated on an integer scale from 0 to 2, yielding a total score ranging from 0 (lowest quality) to 10 (highest quality).

SECONDARY OUTCOMES:
Concordance between photograph-based versus in-person-based diagnosis, as quantified using Cohen's kappa. | 1 hour
  Cohen's kappa is a measure of inter-rater agreement that takes into account the possibility of agreement occurring by chance.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McMahon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connor DM, Jew OS, Perman MJ, Castelo-Soccio LA, Winston FK, McMahon PJ. Diagnostic Accuracy of Pediatric Teledermatology Using Parent-Submitted Photographs: A Randomized Clinical Trial. JAMA Dermatol. 2017 Dec 1;153(12):1243-1248. doi: 10.1001/jamadermatol.2017.4280. PMID 29141082